CLINICAL TRIAL: NCT01861782
Title: Comparison Between Dead Sea Solar and Water Treatment to "Sulfur Pool" and Medicinal Mud Treatment in Patients With Rheumatoid Arthritis
Brief Title: Comparison Between Dead Sea Solar and Water Treatment to Sulfur Pool and Medicinal Mud Treatment in Patients With RA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Mahmoud Abu-Shakra, Head of Rheumatology Clinic, Soroka University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: sor0356-12ctil; 0356-12-SOR (Other: Soroka University Medical Center)
Record Dates: First submitted 2013-05-12; First posted 2013-05-24 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Water Purification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dead Sea Solar and Water Treatment (Experimental): Dead Sea Solar and Water Treatment
  Interventions: Other: Dead Sea Solar and Water Treatment
- Sulfur Pool & Medicinal Mud (Experimental): Sulfur Pool & Medicinal Mud
  Interventions: Other: Sulfur Pool & Medicinal Mud

INTERVENTIONS:
Other: Dead Sea Solar and Water Treatment
  Arms: Dead Sea Solar and Water Treatment
Other: Sulfur Pool & Medicinal Mud
  Arms: Sulfur Pool & Medicinal Mud

SUMMARY:
Prospective open label crossover self controlled study. The study population will randomly be divided into two groups.

The study will take place in Lot Spa Hotel at the Dead Sea in two cycles (one of 16 participants and one of 14 participants) and will be comprised of 3 main stages:

1. Initial exposure to treatment for 14 days excluding Friday and Saturday (each of the two groups will have its own treatment protocol)
2. 12-month washout period
3. Crossover of the two groups and second exposure to treatment for 14 days excluding Friday and Saturday (each of the two groups will have its own treatment protocol).

The population in the study will be composed of patients diagnosed and treated for rheumatoid arthritis at the Soroka University Medical Center who are 18 and above of age.

The patients will be selected by the PI and his team and addressed regarding their willingness to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18
2. Patients with diagnosed rheumatoid arthritis
3. Patients with moderate disease activity (DAS28 > 3.2)

Exclusion Criteria:

1. Patients who suffer from Photosensitivity
2. Patients with Suspected Lupus Erythematoides
3. Patients with tendency to sudden loss of consciousness and/or dizziness
4. Patients under chemotherapeutic treatment
5. Patients with Active Malignancy
6. Patients with lowest level of physical functioning (class 4)
7. Patients with serious uncontrolled concomitant chronic disease
8. Drug Abuser
9. Patients with severe peripheral venous insufficiency
10. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in DAS28 (Disease Activity Score) between the baseline and several occasions after each one of the proposed treatments. | up to 4 months
  DAS28 will be evaluated before and immediately after the treatment, as well as one and 3 months after treatment has started

SECONDARY OUTCOMES:
Assessing the change between baseline and several occasions after each one of proposed the treatments | up to 4 months
  Composite outcome measure : Assessing the change between baseline and several occasions after each one of proposed the treatments by the following parameters:
  * CRP
  * ESR
  * Vitamine D 25 (OH)
  * TNF-α
  * Cytokines (IL1, IL6, IL10, IL17, IL23) The various markers levels will be obtained from serum samples collected before and right after treatment, one month after treatment and 3 months after treatment has started using ELISA method

CONTACTS AND LOCATIONS:
Locations (1):
- Lot Spa Hotel at the Dead Sea, Ein Bokek, Israel